CLINICAL TRIAL: NCT00308906
Title: Assessment of Gene and Urinary Protein Expression in Aminoglycoside-treated and Untreated Infants, Children and Adolescents
Brief Title: Identification of Gene and Protein Markers of Kidney Injury in Aminoglycoside-treated Children
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of Louisville (Other)
Responsible Party: Principal Investigator, Mary Jayne Kennedy, Associate Professor, Virginia Commonwealth University
Other Study IDs: Aminoglycoside Waste Specimen
Record Dates: First submitted 2006-03-29; First posted 2006-03-30 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Infection; Renal Dysfunction
Keywords: infection; renal dysfunction; aminoglycoside; protein; child
MeSH Terms: conditions — Infections; Renal Insufficiency | interventions — Aminoglycosides

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Waste blood samples will be collected in order to evaluate potential genetic mechanisms of aminoglyoside induced renal injury. Waste urine samples will be collected in order to evaluate candidate protein biomarkers of aminoglycoside induced renal injury.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Hospitalized, untreated infants and children
  Interventions: Drug: aminoglycoside
- 2: Aminoglycoside treated infants and children without renal injury
  Interventions: Drug: aminoglycoside
- 3: Aminoglycoside treated infants with renal injury
  Interventions: Drug: aminoglycoside

INTERVENTIONS:
Drug: aminoglycoside — Aminoglycosides will be administered and monitored as part of the routine standard of care for the subject.

SUMMARY:
The purposes of this study are to identify potential gene and protein markers of aminoglycoside-induced kidney injury in infants, children and adolescents treated with aminoglycoside antibiotics.

ELIGIBILITY:
Inclusion Criteria: (1) Hospitalized male and female newborns, infants, children and adolescents (ages birth to 18 years) with a diagnosis of suspected or proven bacterial sepsis, meningitis or other indication necessitating aminoglycoside therapy (2) hospitalized and outpatient newborns, infants, children and adolescents (ages birth to 18 years) who are not receiving aminoglycoside therapy.

Exclusion Criteria: (1) Current treatment with inhaled or ophthalmic aminoglycosides (2) Prior treatment with an aminoglycoside within the last 30 days

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Aminoglycoside treated and untreated newborns, infants and children.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2006-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Indicators of renal injury | Pre and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jayne Kennedy, Pharm.D., Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - University of Lousiville, Louisville, Kentucky
  - Virginia Commonwealth University, Richmond, Virginia